CLINICAL TRIAL: NCT03754790
Title: An Open-label, Long-term Safety and Efficacy Study of Fitusiran in Patients With Hemophilia A or B, With or Without Inhibitory Antibodies to Factor VIII or IX
Brief Title: Long-term Safety and Efficacy Study of Fitusiran in Patients With Hemophilia A or B, With or Without Inhibitory Antibodies to Factor VIII or IX
Acronym: ATLAS-OLE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTE15174; U1111-1210-0018 (Registry Identifier: ICTRP); 2023-508884-59 (Registry Identifier: CTIS); 2018-002880-25 (EudraCT Number)
Record Dates: First submitted 2018-11-25; First posted 2018-11-27 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — fitusiran

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fitusiran (Experimental): Participants will be administered fitusiran as a subcutaneous injection once monthly or every other month for up to 48 months post initiation of modified IMP dose/frequency or until fitusiran becomes commercially available, whichever comes first.
  Interventions: Drug: Fitusiran

INTERVENTIONS:
Drug: Fitusiran — Pharmaceutical form:solution for injection Route of administration: subcutaneous

SUMMARY:
Primary Objective:

To characterize the long-term safety and tolerability of fitusiran

Secondary Objectives:

* To characterize the efficacy and long-term efficacy of fitusiran as assessed by the frequency of:

  * Bleeding episodes
  * Spontaneous bleeding episodes
  * Joint bleeding episodes
* To characterize the effects of fitusiran on health-related quality of life (HRQOL) measures in participants ≥17 years of age

DETAILED DESCRIPTION:
The estimated total time on the study for a participant is up to 90 months (including screening, treatment period and safety follow up period).

ELIGIBILITY:
Inclusion criteria :

* Participant must be at least 12 years of age inclusive, at the time of signing the informed consent
* Participants with severe hemophilia A or B who have completed a Phase 3 fitusiran clinical trial
* Male
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol. In countries where legal age of majority is above 18 years, a specific ICF must also be signed by the participant's legally authorized representative

Exclusion criteria:

* Completion of a surgical procedure within 14 days prior to screening, or currently receiving additional factor concentrate or BPA infusion for postoperative hemostasis
* Current participation in immune tolerance induction treatment (ITI)
* Current use of factor concentrates or bypassing agents (BPAs) as regularly administered prophylaxis designed to prevent spontaneous bleeding episodes except for participants requiring factor concentrates or BPAs prophylaxis during the study dosing pause period
* Use of compounds other than factor concentrates or BPAs for hemophilia treatment
* Current or prior participation in a gene therapy trial
* Alanine aminotransferase (ALT) and/or Aspartate aminotransferase (AST) >1.5 × upper limit of normal reference range (ULN) for patients who are naïve to fitusiran at study start; ALT and/or AST > 5 x ULN for patients who were in the fitusiran arm in the parent study
* Additional exclusions for participants not currently participating in a fitusiran trial at the time of enrollment in the lower dose cohort:

  * Clinically significant liver disease
  * History of arterial or venous thromboembolism

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2026-11-05 (Estimated); Study Completion 2026-11-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events (TEAEs) | from study baseline (day 1) up to maximum 88 months
  The number of participants experiencing any TEAEs, serious TEAEs, discontinuation due to TEAEs and death will be reported

SECONDARY OUTCOMES:
Annualized bleeding rate (ABR) | from first ever dose of fitusiran (day 1) up to maximum 78 months
  Annualized bleeding rate (ABR) in the treatment period
Annualized spontaneous bleeding rate | from first ever dose of fitusiran (day 1) up to maximum 78 months
  Annualized spontaneous bleeding rate in the treatment period
Annualized joint bleeding rate | from first ever dose of fitusiran (day 1) up to maximum 78 months
  Annualized joint bleeding rate in the treatment period
Changes in Haem-A-quality of life (QoL) score | from first ever dose of fitusiran (day 1) up to maximum 78 months
  Change in Haem A QoL physical health score and total score in the treatment period (in participants ≥17 years of age) from first ever dose of fitusiran (day 1) up to maximum 78 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (79):
- United States (10):
  - Phoenix Childrens Hospital Site Number : 8400009, Phoenix, Arizona
  - Children's Hospital Los Angeles Site Number : 8400019, Los Angeles, California
  - Center for Inherited Blood Disorders (CIBD) Site Number : 8400016, Orange, California
  - Nemours Children's Clinic Site Number : 8400008, Jacksonville, Florida
  - St Joseph's Children's Hospital of Tampa Site Number : 8400002, Tampa, Florida
  - Rush University Medical Center -1725 W Harrison St Site Number : 8400001, Chicago, Illinois
  - ~Massachusetts General Hospital Site Number : 8400011, Boston, Massachusetts
  - University of Michigan Hospital - 1500 E Medical Center Dr Site Number : 8400012, Ann Arbor, Michigan
  - Alliance for Childhood Diseases Site Number : 8400007, Las Vegas, Nevada
  - Childrens Hospital Medical Center of Akron Site Number : 8400006, Akron, Ohio
- Australia (3):
  - Investigational Site Number : 0360001, Camperdown, New South Wales
  - Investigational Site Number : 0360003, Prahran, Victoria
  - Investigational Site Number : 0360002, Murdoch, Western Australia
- Investigational Site Number : 1240001, Montreal, Quebec, Canada
- China (13):
  - Investigational Site Number : 1560004, Beijing
  - Investigational Site Number : 1560007, Beijing
  - Investigational Site Number : 1560014, Changsha
  - Investigational Site Number : 1560009, Chengdu
  - Investigational Site Number : 1560002, Guangzhou
  - Investigational Site Number : 1560011, Guiyang
  - Investigational Site Number : 1560005, Hangzhou
  - Investigational Site Number : 1560008, Jinan
  - Investigational Site Number : 1560012, Kunming
  - Investigational Site Number : 1560013, Lanzhou
  - Investigational Site Number : 1560010, Qingdao
  - Investigational Site Number : 1560003, Shanghai
  - Investigational Site Number : 1560006, Suzhou
- Investigational Site Number : 2080001, Copenhagen, Denmark
- France (2):
  - Investigational Site Number : 2500002, Lyon
  - Investigational Site Number : 2500003, Paris
- Germany (2):
  - Investigational Site Number : 2760001, Berlin
  - Investigational Site Number : 2760003, Leipzig
- Investigational Site Number : 3480002, Budapest, Hungary
- India (6):
  - Investigational Site Number : 3560001, Bangalore
  - Investigational Site Number : 3560005, Lucknow
  - Investigational Site Number : 3560007, Mumbai
  - Investigational Site Number : 3560002, Pune
  - Investigational Site Number : 3560010, Pune
  - Investigational Site Number : 3560004, Ranipet
- Ireland (2):
  - Investigational Site Number : 3720001, Crumlin, Dublin
  - Investigational Site Number : 3720002, Dublin
- Investigational Site Number : 3760001, Ramat Gan, Israel
- Italy (2):
  - Investigational Site Number : 3800002, Milan, Lombardy
  - Investigational Site Number : 3800004, Padua, Veneto
- Japan (6):
  - Investigational Site Number : 3920002, Nishinomiya, Hyōgo
  - Investigational Site Number : 3920005, Isehara, Kanagawa
  - Investigational Site Number : 3920003, Kitakyushu
  - Investigational Site Number : 3920001, Nagoya
  - Investigational Site Number : 3920004, Saitama
  - Investigational Site Number : 3920008, Tokyo
- Malaysia (3):
  - Investigational Site Number : 4580003, Ampang
  - Investigational Site Number : 4580001, Johor Bahru
  - Investigational Site Number : 4580002, Kota Kinabalu
- Investigational Site Number : 7100002, Port Elizabeth, South Africa
- South Korea (4):
  - Investigational Site Number : 4100001, Busan, Busan
  - Investigational Site Number : 4100002, Daejeon, Daejeon
  - Investigational Site Number : 4100003, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100004, Seoul
- Taiwan (7):
  - Investigational Site Number : 1580002, Changhua
  - Investigational Site Number : 1580008, Taichung
  - Investigational Site Number : 1580004, Taichung
  - Investigational Site Number : 1580003, Taipei
  - Investigational Site Number : 1580001, Taipei
  - Investigational Site Number : 1580005, Taipei
  - Investigational Site Number : 1580007, Taoyuan
- Turkey (Türkiye) (8):
  - Investigational Site Number : 7920002, Adana
  - Investigational Site Number : 7920004, Akdeniz
  - Investigational Site Number : 7920012, Bornova
  - Investigational Site Number : 7920006, Gaziantep
  - Investigational Site Number : 7920005, Istanbul
  - Investigational Site Number : 7920003, Izmir
  - Investigational Site Number : 7920008, Kayseri
  - Investigational Site Number : 7920007, Samsun
- Ukraine (4):
  - Investigational Site Number : 8040001, Kyiv
  - Investigational Site Number : 8040003, Kyiv
  - Investigational Site Number : 8040002, Lviv
  - Investigational Site Number : 8040004, Mykolaiv
- United Kingdom (2):
  - Investigational Site Number : 8260001, London, London, City of
  - Investigational Site Number : 8260004, Glasgow

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Young G, Kavakli K, Klamroth R, Matsushita T, Peyvandi F, Pipe SW, Rangarajan S, Shen MC, Srivastava A, Sun J, Tran H, You CW, Zulfikar B, Menapace LA, Zhang C, Shen Y, Puurunen M, Demissie M, Kenet G. Safety and efficacy of a fitusiran antithrombin-based dose regimen in people with hemophilia A or B: the ATLAS-OLE study. Blood. 2025 Jun 19;145(25):2966-2977. doi: 10.1182/blood.2024027008. PMID 40053895
- See also: LTE15174 Plain Language Results Summaries — https://www.trialsummaries.com/Study/StudyDetails?id=26149&tenant=MT_SNY_9011